CLINICAL TRIAL: NCT01733472
Title: General Versus Intrathecal Anaesthesia for Patients Undergoing Elective Total Hip Arthroplasty
Brief Title: General or Regional Anesthesia for Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Andreas Harsten, M.D., Region Skane
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hip-CPH-2013; Hässleholm2013 (Other: Region Skåne)
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis
Keywords: anaesthetic techniques; subarachnoid; analgesia
MeSH Terms: conditions — Osteoarthritis; Agnosia | interventions — Remifentanil; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RA-arm (Placebo Comparator): RA-arm: the patients in this arm will receive intrathecal anaesthesia consisting of bupivacaine 15 mg
  Interventions: Drug: RA-arm
- GA-arm, remifentanil (Experimental): GA-arm: patients in this arm will receive general anaesthesia consisting of Target Controlled Infusion (TCI) of remifentanil and propofol
  Interventions: Drug: GA-arm, remifentanil

INTERVENTIONS:
Drug: GA-arm, remifentanil — Remifentanil and propofol will be delivered intravenously via TCI pumps according to the "Marsh" and "Minto" algorithm
  Other Names: GA: TCI consisting of remifentanil an propofol
  Arms: GA-arm, remifentanil
Drug: RA-arm — Intrathecal (i.e. spinal) anesthesia with isobaric bupivacaine 15 mg administered intrathecally at L4-L5.
  Other Names: Regional anesthesia
  Arms: RA-arm

SUMMARY:
The purpose of this study is to determine whether general anaesthesia or regional anaesthesia is best for patients undergoing Total Hip Arthroplasty.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) with a follow up time of 48 hrs. Patients scheduled for primary Total Hip Arthroplasty. A total of 120 patients randomly assigned to one of the two alternatives (general anaesthesia (GA) or regional anaesthesia (RA)).

General anaesthesia compared to intrathecal anaesthesia will give shorter length of hospital stay (LOS) for patients undergoing total hip arthroplasty (THA).

Primary endpoint:

LOS.

Secondary endpoints:

Postoperative pain? Postoperative orthostatic function (dizziness) Time until the patient meets the discharge criteria from PACU How many patients will need at least one urinary bladder catheterisation

ELIGIBILITY:
Inclusion Criteria: patients with osteoarthritis scheduled for surgery

* patients that will require THA
* patients over 45 yrs and under 85 yrs.
* patients that understand the given information and are willing to participate in this study
* patients who have signed the informed consent document.
* patients belonging to ASA class I-III.

Exclusion Criteria:

* prior surgery to the same hip
* patients with a history of stroke, neurological or psychiatric disease that potentially could affect the perception of pain
* obesity (BMI > 35)
* active or suspected infection
* patients taking opioids or steroids
* patients suffering from rheumatoid arthritis or an immunological depression
* patients who are allergic to any of the drugs being used in this study

Ages: 46 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Harsten, M.D., Principal Investigator — Region Skane
Locations (1):
- Dept Orthopedic Surgey, Hässleholm Hospital, PO Box 351,, Hässleholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler SJ, Symons J, Sabato S, Myles PS. Epidural analgesia compared with peripheral nerve blockade after major knee surgery: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2008 Feb;100(2):154-64. doi: 10.1093/bja/aem373. PMID 18211990
- [Background] Marsh BJ, Morton NS, White M, Kenny GN. A computer controlled infusion of propofol for induction and maintenance of anaesthesia in children. Can J Anaesth. 1990 May;37(4 Pt 2):S97. No abstract available. PMID 2361330
- [Background] Minto CF, Schnider TW, Shafer SL. Pharmacokinetics and pharmacodynamics of remifentanil. II. Model application. Anesthesiology. 1997 Jan;86(1):24-33. doi: 10.1097/00000542-199701000-00005. PMID 9009936
- [Background] Harsten A, Kehlet H, Ljung P, Toksvig-Larsen S. Total intravenous general anaesthesia vs. spinal anaesthesia for total hip arthroplasty. Acta Anaesthesiol Scand. 2015 Apr;59(4):542-3. doi: 10.1111/aas.12495. Epub 2015 Mar 3. No abstract available. PMID 25736216

RESULTS

PARTICIPANT FLOW:
Groups:
- RA-arm: RA-arm: the patients in this arm will receive intrathecal anaesthesia consisting of bupivacaine 15 mg
  placebo
Period: Overall Study
Arm/Group | RA-arm | GA-arm, Remifentanil
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RA-arm | GA-arm, Remifentanil | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9) | 66 (8) | 67 (8)
Sex/Gender, Customized [Number; unit: participants]
  Female | 29 | 31 | 60
  Male | 31 | 29 | 60
Region of Enrollment [Number; unit: participants]
  Sweden | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Time from the end of surgery until the patients meets the discharge criteria will be evaluated. Discharge criteria: able to get in and out of bed, Able to get dressed. Able to sit down in a chair and get up again. Able to walk 50 meters wit/without crutches. Able to flex knee 70 degrees. Able to walk stairs. Pain manageable with oral analgesics. Acceptance to be discharged
Time Frame: Up to 4 days after surgery
Population: Two patients in the RA group were excluded because of the conversion to general anaesthesia.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | RA-arm | GA-arm, Remifentanil
Number analyzed (Participants) | 58 | 60
hours | 30 [25 to 45] | 26 [23 to 30]

2. Secondary Outcome: Post Operative Pain
Description: Pain will be monitored using a Visual Analogue Scale. Pain will be monitored with the patient in four different positions. VAS 100 mm used for assessment of pain (0 = no pain, 100 = worst imaginable pain). At each time and position the median VAS-pain score was reported (generally the distribution of pain scores are not normally distributed and hence median value was used)
Time Frame: from end of surgey until 48 hrs later
Population: Two patients in the RA group were excluded because of the conversion to general anaesthesia.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | RA-arm | GA-arm, Remifentanil
Number analyzed (Participants) | 58 | 60
score on a scale | 35 [20 to 50] | 25 [0 to 35]

3. Other Pre Specified Outcome: Time Hrs Until the Patient Meets the Discharge Criteria From PACU
Description: Hours until the patient meets the discharge criteria from PACU will be monitored every 15 min from teh time the patient arrives to PACU until he/she meets the discharge criteria
Time Frame: 12 hrs
Population: Two patients in the RA group were excluded because of the conversion to general anaesthesia.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | RA-arm | GA-arm, Remifentanil
Number analyzed (Participants) | 58 | 60
hours | 4 [3 to 5] | 3 [2 to 4]

ADVERSE EVENTS:
Arm/Group | RA-arm | GA-arm, Remifentanil
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 1/60 | 1/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA-arm (N=60) | GA-arm, Remifentanil (N=60)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) — atrial fibrillation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes